CLINICAL TRIAL: NCT00872092
Title: Validation of Breath Tests in Diagnosing Small Bowel Bacterial Overgrowth
Acronym: BTO
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Heiner K. Berthold, University of Bonn - Germany
Other Study IDs: BTO-0001
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Malabsorption Syndromes
Keywords: small bowel; bacterial overgrowth
MeSH Terms: conditions — Malabsorption Syndromes

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — Breath samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breath test: Subjects with suspected SBBO
  Interventions: Other: Stable-isotope labeled lactose ureide breath test

INTERVENTIONS:
Other: Stable-isotope labeled lactose ureide breath test — 2 g 13C-labeled lactose ureide orally
  Other Names: Lactosyl ureide

SUMMARY:
Normally the gastrointestinal tract is only sparsely colonized with bacteria. The normal flora of the duodenal or jejunal aspirate contains no more than 10^5 bacteria per milliliter. Small bowel bacterial overgrowth (SBBO) is defined as a pathologically increased number of bacteria or the presence of colonic flora in the proximal intestine. The reasons for this condition are manifold, ranging from diabetic neuropathy to surgical bypass. SBBO is frequent in elderly people. Therapy is targeted at correcting the underlying small bowel abnormalities that predispose to the condition and at providing appropriate antibiotic therapy. The symptoms and signs of SBBO can be reversed with this approach. However, in many patients the conditions predisposing to SBBO persist life-long, once present. This suggests that noninvasive, sensitive diagnostic tools with high specificity are required. Bacterial culture of upper intestinal content is considered the diagnostic gold standard. However, since endoscopic harvesting of duodenal or jejunal fluid is difficult and invasive, indirect tests such as breath tests have been advocated as diagnostic tools. Hydrogen breath tests are commonly employed since the substrates can be easily obtained and the measurement is simple. Hydrogen is formed when carbohydrates are fermented in the intestine. Breath hydrogen analysis allows a separation of metabolic activity of the intestinal flora from that of the host, since no known hydrogen production occurs in mammalian tissue. The hydrogen breath test most often used in routine clinical practice uses glucose. However, the utility of this test is mostly limited by its low sensitivity, because there are "nonproducers" in up to 25% of the subjects tested. The investigators have developed a stable isotope breath test using 13C-labeled lactose-ureide. Glycosyl-ureides are condensation products of reducing sugars and urea in aqueous acid. Lactose-[13C]ureide has been used to investigate oro-caecal transit time because it resists digestion by small intestinal enzymes and is hydrolyzed by bacterial enzymes in the large intestine. A number of studies have described the use of this substrate in adults and children. The aim of the present study was to investigate the lactose-[13C]ureide breath test in subjects with suspected SBBO and to compare its results with the results of the glucose hydrogen breath test. Microbiological analyses of upper intestinal bacterial cultures were used as gold standard to identify SBBO.

ELIGIBILITY:
Inclusion Criteria:

* Suspected small bowel bacterial overgrowth

Exclusion Criteria:

* Age < 18 years
* Antibiotic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected small bowel bacterial overgrowth
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 1997-10; Primary Completion 1998-09 (Actual); Study Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
13CO2 enrichment in breath CO2 | 3 hours

SECONDARY OUTCOMES:
Hydrogen output in breath | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Heiner K. Berthold, MD, PhD, Principal Investigator — University of Bonn
Locations (1):
- University of Bonn, Bonn, Germany